CLINICAL TRIAL: NCT02167373
Title: Dashboards for Clinician Monitoring of Patients Through a Mobile Sensing Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cogito Health Inc (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Brigham and Women's Hospital (Other); Partners HealthCare (Other)
Responsible Party: Principal Investigator, Skyler Place, General Manager of Advanced Product Development, Cogito Health Inc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2R44MH100748 (NIH)
Record Dates: First submitted 2014-06-03; First posted 2014-06-19 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Behavioral Health With Medical Comorbidities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental): Cogito Companion Intervention. Participants will be provided with a mobile phone application that provides feedback on their mental health. The participants' clinicians will be provided with a desktop application to review their patients' results.
  Interventions: Other: Cogito Companion Intervention; Device: mobile phone application

INTERVENTIONS:
Other: Cogito Companion Intervention
  Other Names: Cogito Mobile Sensing Platform
  Arms: Intervention
Device: mobile phone application
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether the use of a mobile sensing platform in a primary care setting has an effect on provider workflows, patient outcomes, patient engagement, patient self-help behavior, health research, and total cost of care.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 70 years of age.
* Speak, understand, and read conversational English.
* Be a current patient of South Huntington Clinic recommended for behavioral health care.
* Have a smartphone and cell service plan, including voice and data, that meets the device requirements of the Mobile Sensing Platform.

Exclusion Criteria:

* Planning on permanently leaving Boston during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2015-11; Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Treatment Outcome | Change from baseline to six months later
  Depression will be assessed by the Patient Health Questionnaire-8.
Quality of Life Outcome | Change from baseline to six months later
  Patient reported Schwartz Outcome Scale-10 (SOS-10).

SECONDARY OUTCOMES:
Cost of Care | Measured at six months
  Cost of care can be measured by proxy, through counts of emergency room visits, hospitalization admissions and days, and hospital re-admissions in the last six months.
Patient Engagement | Measured at six months
  Patient engagement will be assessed through frequency of patient use of the mobile technology, no-show rate at appointments, and completion of treatment homework assignments in the last six months.
Self-Help Behavior | Measured at six months
  Self-help behavior will be measured through change in behavior patterns, usage of the mobile application, and requests for additional resources in the last six months.
Clinical Outcome (GAF) | Change from baseline to six months later
  We will use the Global Assessment of Functioning (GAF) to measure overall functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- South Huntington Clinic, Jamaica Plain, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No